CLINICAL TRIAL: NCT02462876
Title: Post-market Study: Evaluation of the GORE® VIABAHN® Endoprosthesis for the Treatment of Popliteal Artery Aneurysm
Brief Title: Evaluation of the GORE® VIABAHN® Endoprosthesis for the Treatment of Popliteal Artery Aneurysm (PAA)
Status: Completed | Type: Observational
Sponsor: W.L.Gore & Associates (Industry)
Responsible Party: Sponsor
Other Study IDs: FPR14-03
Record Dates: First submitted 2015-05-29; First posted 2015-06-04 (Estimated); Results first posted 2020-07-13 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Popliteal Artery Aneurysm
MeSH Terms: conditions — Popliteal Artery Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: GORE® VIABAHN® Endoprosthesis — Treatment of Popliteal Artery Aneurysm with the GORE® VIABAHN® Endoprosthesis.

SUMMARY:
This study will assess the long term safety and performance of the GORE® VIABAHN® Endoprosthesis for the treatment of patients with Popliteal Artery Aneurysms.

ELIGIBILITY:
Inclusion Criteria:

Inclusion to the study requires the patient:

1. Received a GORE® VIABAHN® Endoprosthesis to treat a popliteal artery aneurysm
2. Had a symptomatic aneurysm or asymptomatic aneurysm (≥ 2 cm diameter) of the popliteal artery, or the presence of mural thrombus (< 2 cm) in the popliteal artery;
3. Was 18 years of age or older at the time of the treatment;
4. Had an elective popliteal artery aneurysm procedure;
5. Has provided Informed Consent, personally or through lawful representation as determined by applicable local regulations and state law

Exclusion Criteria:

Prior to or at the time of implant the patient is / has:

1. Bilateral popliteal artery aneurysms with initial treatment on the same day;
2. Thrombotic occlusion of the popliteal artery or PAA;
3. Marfan syndrome or Ehlers-Danlos syndrome;
4. Unable to tolerate antiplatelet therapy;
5. Thrombophilia requiring long term anticoagulation;
6. Known allergies to the GORE® VIABAHN® Endoprosthesis components;
7. Enrolled in another investigational drug or medical device trial where participation may have affected the outcome or treatment of the subject in the popliteal artery aneurysm study with the GORE® VIABAHN® Endoprosthesis or had previous surgery for the popliteal artery aneurysm in the study limb.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a symptomatic aneurysm or asymptomatic aneurysm (≥ 2 cm diameter) of the popliteal artery, or presence of mural thrombus (< 2 cm) in the popliteal artery treated since the date of reimbursement in France.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2020-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nabil Chakfé, Principal Investigator — Hôpitaux Universitaire de Strasbourg
Locations (1):
- Hôpitaux Universitaire de Strasbourg, Strasbourg, France

RESULTS

PARTICIPANT FLOW:
Groups:
- Viabahn: Subjects with popliteal artery aneurysm treated with Gore Viabahn endoprosthesis
Period: Overall Study
Arm/Group | Viabahn
Started | 60
Completed | 33
Not Completed | 27
Not completed — Death | 3
Not completed — Lost to Follow-up | 7
Not completed — Surgical Bypass | 9
Not completed — Amputation Above the Metatarsals | 1
Not completed — 36 months follow-up visit missed | 1
Not completed — Patient did not come back since 4 months follow-up | 1
Not completed — Patient did not come back to the vascular department | 1
Not completed — Patient contacted by phone but never came back for his follow-up visits | 1
Not completed — Patient refused to come back | 1
Not completed — Patient was contacted on Sep 2020. He is fine but refused to come back for his 36 months | 1
Not completed — Patient cancelled the follow-up visit twice time | 1

BASELINE CHARACTERISTICS:
Groups:
- VIABAHN® Endoprosthesis: Subjects with popliteal artery aneurysm treated with Gore Viabahn endoprosthesis
Arm/Group | VIABAHN® Endoprosthesis
Number analyzed (Participants) | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.6 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 58
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  France | 60

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Primary Patency at 12 Months
Description: Primary Patency is defined as blood flow without occlusion maintained through the device after implant without an intervention evaluated at 12 months.
Time Frame: 12 months
Population: Includes all subjects who lost patency within 12 months and all patent subjects with at least a 12 month visit or later.
Measure: Count of Participants; unit: Participants
Arm/Group | Viabahn
Number analyzed (Participants) | 51
Participants
  Patent at 12 Months | 40
  Not Patent | 11

2. Primary Outcome: Number of Subjects With a Safety-related Event at 12 Months
Description: Safety-related events are defined as serious adverse events and adverse events related to the study procedure or the study device through 12 months
Time Frame: 12 months
Population: Includes all subjects who have a serious adverse event or adverse event related to study procedure or device within 12 months and all subjects free from those events with at least a 12 month visit or later.
Measure: Count of Participants; unit: Participants
Arm/Group | Viabahn
Number analyzed (Participants) | 56
Participants
  No Event | 29
  Event(s) | 27

3. Secondary Outcome: Probability of Primary Patency
Description: Primary patency is defined as blood flow without occlusion maintained through the device after implant without an intervention. This outcome is estimated through Kaplan-Meier analysis
Time Frame: 12, 24, and 36 months
Population: All participants are included in the Kaplan-Meier analysis for each time point.
Measure: Number (95% Confidence Interval); unit: probability
Arm/Group | Viabahn
Number analyzed (Participants) | 60
probability
  12 months | 0.795 [0.661 to 0.881]
  24 months | 0.734 [0.592 to 0.834]
  36 months | 0.672 [0.514 to 0.788]

4. Secondary Outcome: Number of Subject With a Safety-related Event at 24 and 36 Months
Description: Safety-related events are defined as serious adverse events and adverse events related to study procedure or study device through 24 and 36 months.
Time Frame: 24 and 36 months
Population: For 24 month outcome, includes all subjects who have a serious adverse event or adverse event related to study procedure or device within 24 months and all subjects free from those events with at least a 24 month visit or later (54 subjects).
  For 36 month outcome, includes all subjects who have a serious adverse event or adverse event related to study procedure or device within 36 months and all subjects free from those events with at least a 36 month visit or later (48 subjects).
Measure: Count of Participants; unit: Participants
Arm/Group | Viabahn
Number analyzed (Participants) | 60
Participants
  24 months: number analyzed (Participants) | 54
  24 months: No Event | 25
  24 months: Event(s) | 29
  36 months: number analyzed (Participants) | 48
  36 months: No Event | 14
  36 months: Event(s) | 34

5. Secondary Outcome: Length of Hospital Stay
Description: The number of days the subject remains in the hospital due to endovascular repair of a popliteal artery aneurysm
Time Frame: During hospitalization, approximately 1-2 days
Measure: Count of Participants; unit: Participants
Arm/Group | Viabahn
Number analyzed (Participants) | 60
Participants
  Days in Hospital = 1 | 28
  Days in Hospital = 2 | 16
  Days in Hospital = 3 | 7
  Days in Hospital = 4 or more | 9

6. Secondary Outcome: Length of Procedure
Description: The number of minutes the subject remains in the operating room or catheterization laboratory due to endovascular repair of a popliteal artery aneurysm.
Time Frame: During procedure, approximately 120 minutes
Population: Subjects with missing procedure times are not included.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Viabahn
Number analyzed (Participants) | 52
minutes | 112.5 (39.0)

7. Secondary Outcome: Probability of Primary Assisted Patency
Description: Primary assisted patency is defined as blood flow maintained through the device after implant regardless of repeat interventions performed (without occlusion). This outcome is estimated through Kaplan-Meier analysis.
Time Frame: 12, 24, and 36 months
Population: All participants are included in the Kaplan-Meier analysis for each time point.
Measure: Number (95% Confidence Interval); unit: probability
Arm/Group | Viabahn
Number analyzed (Participants) | 60
probability
  12 months | 0.814 [0.681 to 0.895]
  24 months | 0.732 [0.589 to 0.832]
  36 months | 0.670 [0.512 to 0.787]

8. Secondary Outcome: Probability of Freedom From Limb Loss
Description: Limb loss is defined as the amputation of the study limb above the metatarsals. This outcome is estimated through Kaplan-Meier analysis.
Time Frame: 12, 24, and 36 months
Population: All participants are included in the Kaplan-Meier analysis for each time point.
Measure: Number (95% Confidence Interval); unit: probability
Arm/Group | Viabahn
Number analyzed (Participants) | 60
probability
  12 months | 0.981 [0.874 to 0.997]
  24 months | 0.981 [0.874 to 0.997]
  36 months | 0.953 [0.821 to 0.988]

9. Secondary Outcome: Probability of Freedom From Repeat Intervention
Description: Repeat Intervention is defined as any endovascular or surgical procedure performed to treat a stenosis or occlusion with the study device(s) or within 5 millimeters of the proximal or distal edge of the device(s), treatment of endoleaks or other reasons. This outcome is estimated through Kaplan-Meier analysis.
Time Frame: 12, 24, and 36 months
Population: All participants are included in the Kaplan-Meier analysis for each time point.
Measure: Number (95% Confidence Interval); unit: probability
Arm/Group | Viabahn
Number analyzed (Participants) | 60
probability
  12 months | 0.788 [0.657 to 0.874]
  24 months | 0.788 [0.657 to 0.874]
  36 months | 0.737 [0.593 to 0.837]

10. Secondary Outcome: Probability of Secondary Patency
Description: Secondary patency is defined as blood flow through the device regardless of repeat interventions performed (with or without occlusion) and freedom from surgical bypass. This outcome is estimated through Kaplan-Meier analysis.
Time Frame: 12, 24, and 36 months
Population: All participants are included in the Kaplan-Meier analysis for each time point.
Measure: Number (95% Confidence Interval); unit: probability
Arm/Group | Viabahn
Number analyzed (Participants) | 60
probability
  12 months | 0.843 [0.711 to 0.918]
  24 months | 0.822 [0.685 to 0.903]
  36 months | 0.791 [0.643 to 0.883]

11. Secondary Outcome: Number of Subjects With Technical Success
Description: Technical success is defined as successful aneurysmal exclusion using the study device at time of the procedure without Type I or III endoleaks that require post-procedure intervention within 30 days.
Time Frame: Post-procedure at day 30
Population: Subjects who are not technical failures must have at least 31 days of follow-up in order to be considered a technical success.
Measure: Count of Participants; unit: Participants
Arm/Group | Viabahn
Number analyzed (Participants) | 58
Participants
  Success | 57
  Failure | 1

ADVERSE EVENTS:
Time Frame: 36 months
Arm/Group | VIABAHN® Endoprosthesis
All-Cause Mortality (participants affected / at risk) | 3/60
Serious Adverse Events (participants affected / at risk) | 32/60
Other Adverse Events (participants affected / at risk) | 0/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VIABAHN® Endoprosthesis (N=60)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Anemia iron deficiency (Blood and lymphatic system disorders) | 1 (1)
Cardiac failure Nitric Oxide Synthases (NOS) (Cardiac disorders) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1)
Coronaropathy (Cardiac disorders) | 1 (1)
Death (General disorders) | 2 (2)
Endoleak (General disorders) | 1 (2)
Oedema peripheral (General disorders) | 1 (1)
Vascular stent thrombosis (General disorders) | 1 (2)
Postoperative wound infection (Infections and infestations) | 1 (1)
Renal cyst infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 2 (2)
Sinus infection (Infections and infestations) | 1 (1)
False aneurysm (Injury, poisoning and procedural complications) | 1 (1)
Peripheral artery restenosis (Injury, poisoning and procedural complications) | 1 (1)
Pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1)
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Pancreatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Thrombosis in device (Product Issues) | 5 (6)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory insufficiency (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Ankle ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Aneurysm repair (Surgical and medical procedures) | 1 (2)
Coronary Artery Bypass Graft (CABG) (Surgical and medical procedures) | 1 (1)
Femoral-tibial arterial bypass (Surgical and medical procedures) | 1 (1)
Femoropopliteal artery bypass (Surgical and medical procedures) | 1 (1)
Nephrectomy (Surgical and medical procedures) | 1 (1)
Abdominal aneurysm (Vascular disorders) | 1 (1)
Abdominal aneurysm, ruptured (Vascular disorders) | 1 (1)
Abdominal aortic aneurysm (Vascular disorders) | 1 (1)
Aneurysm enlargement (Vascular disorders) | 1 (1)
Arteriovenous fistula (Vascular disorders) | 1 (1)
Claudication (Vascular disorders) | 1 (1)
Femoral artery aneurysm (Vascular disorders) | 1 (1)
Femoral artery thrombosis (Vascular disorders) | 1 (1)
Hematoma (Vascular disorders) | 1 (1)
Iliac artery stenosis (Vascular disorders) | 1 (1)
Intermittent claudication (Vascular disorders) | 1 (1)
Ischaemic limb pain (Vascular disorders) | 1 (1)
Ischemia (Vascular disorders) | 1 (1)
Ischemia peripheral (Vascular disorders) | 1 (1)
Ischemic limb pain (Vascular disorders) | 1 (1)
Leg ischemia (Vascular disorders) | 2 (2)
Peripheral artery aneurysm (Vascular disorders) | 2 (2)
Peripheral ischaemia (Vascular disorders) | 2 (2)
Popliteal artery aneurysm (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2015-07-14): https://cdn.clinicaltrials.gov/large-docs/76/NCT02462876/Prot_000.pdf
  • Statistical Analysis Plan (2016-07-22): https://cdn.clinicaltrials.gov/large-docs/76/NCT02462876/SAP_001.pdf